CLINICAL TRIAL: NCT05307601
Title: Evaluation of the Cytokine 's Profile Following SarsCov 2 Infection (COVID-19) in Hemodialysis Patients
Brief Title: Immune Response Following COVID-19 in Hemodialysis Patients
Acronym: IMMUNOVIDIAL
Status: Completed | Type: Observational
Sponsor: AURA Paris (Other)
Responsible Party: Sponsor
Other Study IDs: 2020-A01426-33
Record Dates: First submitted 2022-03-24; First posted 2022-04-01 (Actual); Last update posted 2022-04-01 (Actual); Status verified 2022-03

CONDITIONS: Dialysis; Complications; COVID-19; Cytokine Storm
Keywords: dialysis; cytokine; COVID-19
MeSH Terms: conditions — COVID-19; Cytokine Release Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Patients with chronic kidney disease (CKD), particularly those undergoing hemodialysis (HD), are at high risk of a severe form of COVID-19.

This study aims to characterize the inflammatory and antiviral response during SarsCov2 infection in adult

DETAILED DESCRIPTION:
Inclusion criteria were (1) Adult (>18 years old) patient on HD > 6 months, and (2) infection by SARS-CoV-2. Diagnosis of COVID-19 was assessed by Reverse-Transcriptase-Polymerase Chain Reaction (RT-PCR) for SARS-CoV-2 in nasopharyngeal swab or by typical COVID-19 radiological images on thoracic computerized tomography (CT scan).

Severe forms of COVID-19 were defined as requiring oxygen therapy, admission in intensive care unit (ICU) or death

Primary end point :

* Characterization the cytokine's profile at the early (day 7) and inflammatory (day 14) phase of COViD-19 in HD patient

Secondary End points :

* Analyse the kinetic of the antiviral response (type I and III interferon ) between the early (day 7) and inflammatory (day 14) phase of COViD-19.
* Analyse the kinetic of proinflammatory cytokine response between the early (day 7) and inflammatory (day 14) phase of COViD-19.
* Define an antiviral signature associated with severe form of COVID-19
* Define an anti inflammatory signature associated with severe form of COVID-19

Cytokine's profile is define by the measure of 28 cytokines by Luminex technology

ELIGIBILITY:
Inclusion Criteria:

* Adult (>18 years old) patient on HD > 6 months, and
* Infection by SARS-CoV-2. Diagnosis of COVID-19 was assessed by Reverse-Transcriptase-Polymerase Chain Reaction (RT-PCR) for SARS-CoV-2 in nasopharyngeal swab or by typical COVID-19 radiological images on thoracic computerized tomography (CT scan). The date of diagnosis was defined as the day when RT-PCR or CT-scan confirmed the diagnosis.

Exclusion Criteria:

* Inability to give consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult HD patients from 2 main dialysis units of the AURA: AURA Paris Plaisance and Saint-Ouen
Sampling Method: Non-Probability Sample
Enrollment: 21 (Actual)
Dates: Start 2020-09-01 (Actual); Primary Completion 2021-09-01 (Actual); Study Completion 2021-10-30 (Actual)

PRIMARY OUTCOMES:
Characterization of the cytokine profile during the early phase of COVID-19 | Measurement at Day 7 of COVID-19
  Measurement of 29 cytokines by Luminex including type I and Type III Interferon
Characterization of the cytokine profile during the inflammatory phase of COVID-19 | Measurement at Day 14 of COVID-19]
  Measurement of 29 cytokines by Luminex including type I and Type III Interferon

CONTACTS AND LOCATIONS:
Overall Officials: Maxime Touzot, MD, PhD, Principal Investigator — AURA Paris
Locations (1):
- AURA Paris, Paris, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mutinelli-Szymanski P, Hude I, Merle E, Lombardi Y, Seris P, Abtahi M, Azeroual L, Bourgain C, Ensergueix G, Katerinis I, Kolko A, Kolta A, Maheas C, Mehrbanian S, Morel P, Ossman R, de Preneuf H, Roux A, Saltiel C, Vende F, Verhoeven AS, Viron B, Laplanche S, Le Monnier A, Ridel C, Urena-Torres P, Touzot M. Neutrophil:lymphocyte ratio predicts short-term outcome of COVID-19 in haemodialysis patients. Clin Kidney J. 2020 Nov 21;14(1):124-131. doi: 10.1093/ckj/sfaa194. eCollection 2021 Jan. PMID 33558835
- [Background] Pedersen SF, Ho YC. SARS-CoV-2: a storm is raging. J Clin Invest. 2020 May 1;130(5):2202-2205. doi: 10.1172/JCI137647. PMID 32217834
- [Background] Kato S, Chmielewski M, Honda H, Pecoits-Filho R, Matsuo S, Yuzawa Y, Tranaeus A, Stenvinkel P, Lindholm B. Aspects of immune dysfunction in end-stage renal disease. Clin J Am Soc Nephrol. 2008 Sep;3(5):1526-33. doi: 10.2215/CJN.00950208. Epub 2008 Aug 13. PMID 18701615
- [Background] Chen G, Wu D, Guo W, Cao Y, Huang D, Wang H, Wang T, Zhang X, Chen H, Yu H, Zhang X, Zhang M, Wu S, Song J, Chen T, Han M, Li S, Luo X, Zhao J, Ning Q. Clinical and immunological features of severe and moderate coronavirus disease 2019. J Clin Invest. 2020 May 1;130(5):2620-2629. doi: 10.1172/JCI137244. PMID 32217835